CLINICAL TRIAL: NCT05489822
Title: Sponsor-initiated, Prospective, Single-center, Non-interventional Clinical Observational Study to Evaluate the VERTICALE® Cervical System in Spine Surgery According to Its Intended Use.
Brief Title: PMCF Study to Evaluate the VERTICALE® Cervical System in Spine Surgery According to Its Intended Use.
Status: Recruiting | Type: Observational
Sponsor: Silony Medical GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: TDII_2014-003_2.1_103
Record Dates: First submitted 2022-07-27; First posted 2022-08-05 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Degenerative Disc Disease (DDD); Instabilities; Trauma; Deformity
Keywords: NDI
MeSH Terms: conditions — Intervertebral Disc Degeneration; Wounds and Injuries; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: VERTICALE® Cervical System — All measures and devices mentioned in the study protocol correspond to routine clinical practice with the exception of the following questionnaires:
  NDI (Neck Disability Index) NRS (Numerical Rating Scale) neck pain (cervical spine) and NRS arm pain mJOA (modified Japanese Orthopaedic Association) Score

SUMMARY:
In accordance with the European Medical Device Regulation MDR 2017/745/EU, the legal manufacturers of medical devices are obliged to evaluate medical devices with regard to their clinical performance and safety.

The VERTICALE® Cervical System is intended for immobilization and stabilization of spinal segments of the craniocervical junction (occipital-C2), subaxial cervical spine (C3-C7) and upper thoracic spine (T1-T3).

Primary Objective:

To assess the functional outcome and clinical benefit of the VERTICALE® Cervical System for the patient using the NDI (Neck Disability Index) questionnaire.

Primary endpoint hypothesis:

The investigators hypothesize that NDI improves by at least 10% or 5 points at 12 months FU (Follow-Up) compared with preoperatively.

DETAILED DESCRIPTION:
In accordance with the European Medical Device Regulation MDR 2017/745/EU, the legal manufacturers of medical devices are obliged to evaluate medical devices with regard to their clinical performance and safety.

The VERTICALE® Cervical System is intended for immobilization and stabilization of spinal segments of the craniocervical junction (occipital-C2), subaxial cervical spine (C3-C7) and upper thoracic spine (T1-T3).

The investigators interest is the continuous improvement of the surgical procedure in the context of degenerative cervical spine diseases. Patient satisfaction, as well as the avoidance of possible complications, are the main focus here. In addition, CE-certified medical devices must be evaluated for long-term performance and safety in clinical practice in accordance with the Medical Devices Act. The VERTICALE® Cervical System is a rod-screw system for immobilization (= immobilization) and stabilization of the affected segments, in the area between the occiput, the cervical spine and the upper thoracic spine (up to the 3rd thoracic vertebral body). Surgical intervention with the VERTICALE® Cervical System is performed from behind (posteriorly) and usually serves to stiffen the affected areas.

The goals of surgical intervention depend on the exact clinical picture and the associated symptoms, but usually consist of surgical relief of the affected structures of the nervous apparatus and/or spinal cord, stabilization of the bony structures to restore and/or maintain function, and relief of pain.

ELIGIBILITY:
Inclusion Criteria:

Ability to read, understand and speak the local language fluently to ensure understanding of Informed consent and protocol specific investigations

* The surgical indication must be one or a combination of the following
* Degenerative disc disease (DDD)
* Instabilities
* Trauma
* Deformities
* Mono-, bi- and multisegmental restoration (occipital T3)
* Age: ≥ 18 years
* The subject must give written informed consent before inclusion into the PMCF study.

Exclusion Criteria:

Relative and absolute contraindications according to IFU (Instruction for Use):

Under certain circumstances, implantation is prohibited or associated with substantial risks, even though there may be an indication for it.

These include in particular:

* Anticipated or documented allergy or intolerance to the materials (e.g., titanium or cobalt chromium).
* Active systemic infection or an infection localized to the site of the proposed implantation
* Any case in which the chosen implants would be too large or too small to achieve a successful result.
* Any patient for whom the use of the implant would conflict with anatomical structures.
* Missing bony structures, which would render solid anchoring of the implant impossible (e.g., in the case of fractures, tumors, or osteoporosis). In addition, the patient's occupation or activity level or mental capacity may be relative contraindications to this surgery. Specifically, patients who because of their occupation or lifestyle, drug abuse, may place undue stresses on the implant during bony healing and may be at higher risk for implant failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (minimum 18 years old) who undergo surgery with the VERTICALE® Cervical System due to one or a combination of the above mentioned indications and give their written consent to participate.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change of Neck Disability Index (NDI) preoperative (pre-op) compared to 3 month (± 1 month) and 12 months follow-up (± 1 month) | pre-op compared to 3 month (± 1 month) and 12 months follow-up (± 1 month)
  The primary endpoint for this PMCF (Post-Market Clinical Follow-Up) study will be the PROM (Patient-reported Outcome Measurement) instrument Neck Disability Index (NDI). This questionnaire is scientifically accepted. [1] The aim is to show an improvement of the NDI in comparison pre-op to post-op (12 months follow-up (± 1 month)). The reference for the primary endpoint NDI is a 2008 publication by Hovard Vernon, "The Neck Disability Index: State-of-the-Art, 1991-2008." [1] This comparative overview is referenced several times in other publications and represents the SoTA.

SECONDARY OUTCOMES:
Documentation of Complications | intra-op
  Documentation of Complications if any occurred incl. classification in relation to implant and manifestation
Documentation of Complications | Hospital discharge
  Documentation of Complications if any occurred incl. classification in relation to implant and manifestation
Documentation of Complications | 3 month (± 1 month)
  Documentation of Complications if any occurred incl. classification in relation to implant and manifestation
Documentation of Complications | 12 months follow-up (± 1 month)
  Documentation of Complications if any occurred incl. classification in relation to implant and manifestation
Examination of clinical performance | pre-op
  Evaluation by means of X-ray images and, if necessary, supplementary sectional imaging (CT or MRT)
Examination of clinical performance | 3 month (± 1 month)
  Evaluation by means of X-ray images and, if necessary, supplementary sectional imaging (CT or MRT)
Examination of clinical performance | optional: 12 months follow-up (± 1 month))
  Evaluation by means of X-ray images and, if necessary, supplementary sectional imaging (CT or MRT)
Device effectiveness/patient satisfaction: Change of arm/shoulder pain using a Numerical Rating Scale | pre-op compared to post-op (3 month (± 1 month) and 12 months follow-up (± 1 month))
  Documentation of change in pain measured with theNumerical Rating Scale for arm/shoulder pain (0 = no pain; 10 = Unbearable pain).
Device effectiveness/patient satisfaction: Change of neck pain using a Numerical Rating Scale | pre-op compared to post-op (3 month (± 1 month) and 12 months follow-up (± 1 month))
  Documentation of change in pain measured with the Numerical Rating Scale for neck pain (0 = no pain; 10 = Unbearable pain).
Device effectiveness/patient satisfaction: modified Japanese Orthopaedic Association (mJOA) score for the assessment of a possibly present myelopathy. | pre-op
  Acquisition of the mJOA score for the assessment of a possibly present myelopathy. (Range 0-18 Points; 18 points = no myelopathy; 15-17 points = mild myeolopathy; 12-14 points = moderate myelopathy; 0-11 Points = severe myelopathy;
Device effectiveness/patient satisfaction: modified Japanese Orthopaedic Association (mJOA) score for the assessment of a possibly present myelopathy. | 3 month (± 1 month) and 12 months follow-up (± 1 month)
  Acquisition of the mJOA score for the assessment of a possibly present myelopathy. (Range 0-18 Points; 18 points = no myelopathy; 15-17 points = mild myeolopathy; 12-14 points = moderate myelopathy; 0-11 Points = severe myelopathy;
Device effectiveness/patient satisfaction: modified Japanese Orthopaedic Association (mJOA) score for the assessment of a possibly present myelopathy. | 12 months follow-up (± 1 month)
  Acquisition of the mJOA score for the assessment of a possibly present myelopathy. (Range 0-18 Points; 18 points = no myelopathy; 15-17 points = mild myeolopathy; 12-14 points = moderate myelopathy; 0-11 Points = severe myelopathy;

CONTACTS AND LOCATIONS:
Overall Officials: Ankit I. Mehta, MD, Principal Investigator — University of Illinois Hospital and Health Sciences System - UI Health
Locations (1):
- University of Illinois Hospital and Health Sciences System - UI Health, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vernon H. The Neck Disability Index: state-of-the-art, 1991-2008. J Manipulative Physiol Ther. 2008 Sep;31(7):491-502. doi: 10.1016/j.jmpt.2008.08.006. PMID 18803999
- [Background] Kato S, Oshima Y, Oka H, Chikuda H, Takeshita Y, Miyoshi K, Kawamura N, Masuda K, Kunogi J, Okazaki R, Azuma S, Hara N, Tanaka S, Takeshita K. Comparison of the Japanese Orthopaedic Association (JOA) score and modified JOA (mJOA) score for the assessment of cervical myelopathy: a multicenter observational study. PLoS One. 2015 Apr 2;10(4):e0123022. doi: 10.1371/journal.pone.0123022. eCollection 2015. PMID 25837285